CLINICAL TRIAL: NCT03688334
Title: Acute Effects of Oxygen Supplementation During Exercise Among Patients With Idiopathic Pulmonary Fibrosis Without Resting Hypoxemia
Brief Title: Acute Effects of Oxygen Supplementation Among IPF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Afroditi Boutou, Consultant in Respiratory Medicine, George Papanicolaou Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 804/2018
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPF patients (Active Comparator): Supplementation of oxygen treatment (40% FiO2) during steady state cardiopulmonary exercise testing
  Interventions: Drug: Oxygen 40 %
- IPF patients (crossover) (Sham Comparator): Supplementation of medical air (sham Oxygen) during steady state cardiopulmonary exercise testing
  Interventions: Drug: Medical air (sham O2)

INTERVENTIONS:
Drug: Oxygen 40 % — Oxygen supplementation (40%) via Venturi mask
  Arms: IPF patients
Drug: Medical air (sham O2) — Medical air supplementation via Venturi mask
  Arms: IPF patients (crossover)

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a disease characterised with significant morbidity and poor prognosis. Dyspnoea and impaired exercise capacity are very common manifestations of the disease, and result in significant impairment of patients' quality of life. Although hypoxemia is common among subjects with IPF, published data on the effects of supplementary oxygen therapy on specific clinical outcomes among these patients are currently few, while the existing data on the potential benefits of oxygen supplementation to treat exercise-induced hypoxemia, in this patient population, are even more controversial.

Based on the aforementioned, the purpose of this prospective, cross-over clinical trial is to investigate the acute effects of supplemental oxygen administration on the: a) exercise capacity, b) severity of dyspnea, c) cerebral oxygenation, b) muscle oxygenation, and e) hemodynamic profile, as compared to delivery of medical air (sham oxygen), in a group of patients with IPF, without resting hypoxemia, during steady state cardiopulmonary exercise testing (CPET).

ELIGIBILITY:
Inclusion Criteria:

Stable IPF patients with no hospitalization, exacerbation or change in regular IPF medication during the last month, who do not present with resting hypoxemia, but manifest exercise induced hypoxemia

Exclusion Criteria:

1. Major contraindications for CPET conduction
2. Not provision of informed consent -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Exercise duration | through study completion, an average of a year
  Exercise duration (minutes) of steady state cardiopulmonary exercise testing until exhaustion

SECONDARY OUTCOMES:
Dyspnea | through study completion, an average of a year
  maximum dyspnea assessed with modified Borg dyspnea scale (range from 0: nothing at all to 10: maximum dyspnea), during steady state cardiopulmonary exercise testing
Fatigue | through study completion, an average of a year
  maximum fatigue assessed by Borg's Rating of Perceived Exertion Scale (range from 6: no exertion to 20: maximal exertion), during steady state cardiopulmonary exercise testing

OTHER OUTCOMES:
Cerebral oxygenated hemoglobin | through study completion, an average of a year
  The minimum value of cerebral oxygenated hemoglobin during steady state cardiopulmonary exercise testing
Cardiac output | through study completion, an average of a year
  The maximum value of cardiac output in L/min during steady state cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini Markopoulou, MD, PhD, Study Chair — "G. Papanikolaou" General Hospital, Thessaloniki, Greece
Locations (1):
- "G. Papanikolaou" General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No